CLINICAL TRIAL: NCT06980285
Title: ACL Reconstruction With Quadriceps Tendon Graft vs. Quadrupled Semitendinosus Graft: A Comparison of Patients From the Danish National ACL Reconstruction Database
Brief Title: Comparison of Quadriceps and Semitendinosus Grafts in ACL Reconstruction Using Data From the Danish Knee Ligament Reconstruction Registry (DKRR)
Status: Not yet recruiting | Type: Observational
Sponsor: Abdirahman Hassan Omar (Other)
Collaborators: Søernes Privathospital (Other)
Responsible Party: Sponsor-Investigator, Abdirahman Hassan Omar, Medical student, Principal incestigator, Søernes Privathospital
Organization: Søernes Privathospital (Other)
Other Study IDs: SOPH-ACL-3+25
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Anterior Cruciate Ligament Injury; Knee Injury; Ligament Reconstruction; Sports Injuries
Keywords: ACL reconstruction; Quadriceps tendon graft; Semitendinosus graft; DKRR; Knee ligament injury; Orthopaedic surgery; Registry study
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Quadriceps tendon graft: Patients who underwent primary ACL reconstruction using a quadriceps tendon autograft, with or without a bone block. Data are derived retrospectively from the Danish Knee Ligament Reconstruction Registry (DKRR).
- Semitendinosus graft: Patients who underwent primary ACL reconstruction using a quadrupled semitendinosus tendon autograft. Data are derived retrospectively from the Danish Knee Ligament Reconstruction Registry (DKRR).

SUMMARY:
This study looks at two different types of tendon (tissue) used in knee surgery to repair a torn anterior cruciate ligament (ACL), which is a common injury in active people. The two types are taken from different muscles in the thigh: one from the front (quadriceps) and one from the back (semitendinosus). We will use information already collected in a national health registry to see how patients recover after surgery. The study will compare knee function, activity level, and how often patients need another operation.

DETAILED DESCRIPTION:
This is a retrospective observational cohort study based on data from the Danish Knee Ligament Reconstruction Registry (DKRR). The study includes patients who underwent primary ACL reconstruction using either a quadriceps tendon graft (with or without a bone block) or a quadrupled semitendinosus tendon graft. The primary outcome measures are the Knee Injury and Osteoarthritis Outcome Score (KOOS) and the Tegner Activity Scale. Secondary outcomes include reoperation rates, postoperative complications, and patient satisfaction. All available demographic, operative, and patient-reported outcome data will be analyzed. Multivariable regression will be used to adjust for confounders such as age, sex, BMI, time from injury to surgery, and surgeon volume. The study is exempt from ethical approval under Danish law, and data will be handled in compliance with GDPR.

ELIGIBILITY:
Inclusion Criteria:

* Primary ACL reconstruction registered in the Danish Knee Ligament Reconstruction Registry (DKRR)
* Known graft type: quadriceps tendon or semitendinosus tendon Minimum 1-year follow-up with completed patient-reported outcome measures (KOOS and/or Tegner score)
* Age between 15 and 50 years at the time of surgery (optional subgroup analysis)

Exclusion Criteria:

* Revision ACL reconstruction
* Multiligament knee reconstruction
* Missing or incomplete PROMs or key clinical data

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients registered in the Danish Knee Ligament Reconstruction Registry (DKRR) who underwent primary anterior cruciate ligament reconstruction using either a quadriceps tendon graft or a semitendinosus tendon graft. All included patients have completed at least one year of follow-up and patient-reported outcome measures. The population consists of physically active individuals aged 15 to 50 years.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The Knee Injury and Osteoarthritis Outcome Score (KOOS) | At minimum 1 year follow up postoperatively
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) evaluates pain, symptoms, daily living, sport/recreation, and knee-related quality of life.
  Metric type: continuous PROM-based subscale score Method of measurement: Self reported questionnaire
Tegner Activity Score | Minimum 1 year follow up postoperatively.
  Assesses patients' level of physical activity before injury and at follow-up.
  Metric type: Scale from 0-10, where 0 is no physical activity caused by knee problems and 10 is an ability to compete in elite level sport like soccer and ski.
  Method of measurement: Tegner scale, self reported

SECONDARY OUTCOMES:
Re-operation rate | Within 1 year of surgery
  Incidence of surgical re-intervention after primary ACL reconstruction. Method of measurement: Registry recorded re-operations in DKRR
Postoperative complications | Within 1 year after surgery
  Frequency of postoperative complications such as infection, stiffness, or graft failure.
  Metric type: Occurrence of postoperative complications Method of measurement: Clinically reported and registry documented complications in DKRR
Patient satisfaction | 1 year follow up
  Overall patient satisfaction with surgical outcome, if available in registry. Metric type: PROM's available from the DKRR Method of measurement: Patient reported satisfaction score.

CONTACTS AND LOCATIONS:
Locations (1):
- Søernes Privathospital, Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided